CLINICAL TRIAL: NCT04959903
Title: A Phase I/II Study Evaluating the Safety and the Efficacy of SMART101 Injection to Accelerate Immune Reconstitution After T Cell Depleted Allogeneic Hematopoietic Stem Cell Transplantation in Pediatric and Adult Patients With Hematological Malignancies
Brief Title: Safety and Efficacy of SMART101 in Pediatric and Adult Patients With Hematological Malignancies After T Cell Depleted Allo-HSCT
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Smart Immune SAS (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SI101-01
Record Dates: First submitted 2021-07-01; First posted 2021-07-13 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Hematological Malignancies
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Adult patients affected by hematological malignancies (Experimental): Adult patients affected by acute leukemia (AML, ALL or acute leukemia of ambiguous lineage) or myelodysplastic syndrome eligible for a T depleted allogeneic HSCT
  Interventions: Biological: Allogeneic T cell progenitors, cultured ex-vivo
- Pediatric patients affected by hematological malignancies (Experimental): Pediatric patients affected by acute leukemia (AML, ALL or acute leukemia of ambiguous lineage) eligible for a T depleted allogeneic HSCT
  Interventions: Biological: Allogeneic T cell progenitors, cultured ex-vivo

INTERVENTIONS:
Biological: Allogeneic T cell progenitors, cultured ex-vivo — Injection of T cell progenitors at [Day 4-Day 10] after T cell depleted allogeneic HSCT
  Other Names: SMART101

SUMMARY:
The purpose of this study is to evaluate the safety and the efficacy of SMART101 (Human T Lymphoid Progenitor (HTLP)) injection to accelerate immune reconstitution after T cell depleted allogeneic hematopoietic stem cell transplantation (HSCT) in adult and pediatric patients with hematological malignancies.

ELIGIBILITY:
Inclusion Criteria:

Group A (adults):

1. Adult patients affected by:

   * Acute leukemia (AML, ALL) defined as:

     * Acute Myeloid Leukemia (AML):

       * High risk AML in CR1; any adverse genetic abnormality, secondary or therapy related AML excluding good risk genetic abnormalities
       * Chemo-refractory relapse (MRD+)
       * ≥ CR2
     * Acute Lymphoblastic Leukemia (ALL):

       * Chemo-refractory relapse (MRD+)
       * High risk ALL in CR1; Philadelphia (like) or any poor risk feature
       * ≥ CR2
     * Acute leukemia of ambiguous lineage:

       * ≥ CR1 with a minimal residual disease (MRD) <5% (flow cytometry, molecular and/or cytogenetics accepted)
   * Myelodysplastic Syndrome (MDS) with least one of the following:

     * Revised International Prognostic Scoring System risk score of intermediate or higher at the time of transplant evaluation.
     * Life-threatening cytopenia.
     * Karyotype or genomic changes that indicate high risk for progression to acute myelogenous leukemia, including abnormalities of chromosome 7 or 3, mutations of TP53, or complex or monosomal karyotype.
     * Therapy related disease or disease evolving from other malignant processes.
2. Patient eligible for a T-depleted allogeneic HSCT
3. Age ≥ 18y and clinical condition compatible with allogeneic stem cell transplantation
4. Karnofsky index ≥ 70% prior to conditioning regimen
5. Patients with normal organ function prior to conditioning regimen

Group B (pediatrics):

1. Pediatric patients affected by acute leukemia defined as:

   * Acute Myeloid Leukemia (AML):

     * High risk AML in CR1; any adverse genetic abnormality, secondary or therapy related AML excluding good risk genetic abnormalities,
     * Chemo-refractory relapse (MRD+)
     * ≥ CR2
   * Acute Lymphoblastic Leukemia (ALL):

     * Chemo-refractory relapse (MRD+)
     * High risk ALL in CR1; Philadelphia (like) or any poor risk feature
     * ≥ CR2
   * Acute leukemia of ambiguous lineage:

     * ≥ CR1 with a minimal residual disease (MRD) <5% (flow cytometry, molecular and/or cytogenetics accepted)
2. Patient eligible for a T-depleted allogeneic HSCT
3. Age < 18y at the time of inclusion
4. Absence of a matched sibling donor (MSD)
5. Lansky ≥ 70% / Karnofsky performance status ≥ 70% prior to conditioning regimen
6. Patients with normal organ function prior to conditioning regimen

Exclusion Criteria:

Groups A and B:

1. Use of an HLA matched Cord Blood (8/8 allele matched) or haploidentical donor
2. Prior therapy with allogeneic stem cell transplantation
3. Treatment with another cellular therapy within one month before inclusion

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-03-31 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of grade III-IV GvHD | 100 days post-HSCT
  to evaluate the safety profile of the study drug
Occurrence of adverse events related to SMART101 | 100 days post-HSCT
  Number of adverse events and serious adverse events related to SMART101 tabulated for each dose and by age group to evaluate the safety profile of the study drug
CD4+ T cell count | 100 days post-HSCT
  to evaluate the efficacy of the study drug

SECONDARY OUTCOMES:
T cell immune reconstitution | up to Month 12 post-HSCT
  Time course of the T cell immune reconstitution, with a focus on naive CD4+ cells and total CD8+ cells
Cumulative incidence of infections | Day 90, and Months 6, 12 and 24 post-HSCT
Non-relapse mortality (NRM) | Day 90, and Months 6, 12 and 24 post-HSCT

OTHER OUTCOMES:
Overall Survival (OS) | Month 24 post-HSCT
Disease-free Survival | Month 24 post-HSCT

CONTACTS AND LOCATIONS:
Overall Officials: Jaap-Jan BOELENS, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center (MSKCC)
Locations (1):
- Memorial Sloan Kettering Cancer Center (MSKCC), New York, New York, United States

IPD SHARING:
Plan to Share IPD: No